CLINICAL TRIAL: NCT06064916
Title: Visual Outcomes and Patient Satisfaction With Vivity IOL in Post Refractive Patients
Status: Completed | Type: Observational
Sponsor: Berkeley Eye Center (Other)
Responsible Party: Sponsor
Other Study IDs: 69865263
Record Dates: First submitted 2023-09-12; First posted 2023-10-03 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pseudophakia
Keywords: Vivity; Pseudophakia
MeSH Terms: conditions — Pseudophakia | interventions — Visual Acuity; Surveys and Questionnaires; Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Vivity IOL Group: Patients with bilateral implantation of Vivity IOLs.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Defocus Curve; Other: Intraocular Lens Satisfaction (IOLSAT) Questionnaire; Other: Quality of Vision After Surgery (QUVID) Questionnaire; Other: Visual Disturbance Questionnaire; Diagnostic Test: Topography and Tomography

INTERVENTIONS:
Diagnostic Test: Visual Acuity — Monocular and binocular measurement of distance, intermediate, and near visual acuity
Diagnostic Test: Defocus Curve — Measurement of a defocus curve
Other: Intraocular Lens Satisfaction (IOLSAT) Questionnaire — Self-reported post-operative patient satisfaction with vision after surgery
Other: Quality of Vision After Surgery (QUVID) Questionnaire — Self-reported post-operative patient vision quality after surgery
Other: Visual Disturbance Questionnaire — Questionnaire of self-reported visual disturbances of patients
Diagnostic Test: Topography and Tomography — Topography and tomography measurements with Atlas, iTrace, and/or Pentacam

SUMMARY:
This is a non-interventional, prospective, observational study of the outcomes for post myopic refractive surgery patients following successful, uncomplicated cataract surgery with bilateral implantation of the Vivity IOL (DAT***/CCWET*).

Patients will be assessed for monocular and binocular distance, intermediate, and near vision.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, single center, bilateral, observational study of the outcomes for 40 post myopic refractive surgery patients following successful, uncomplicated cataract surgery with bilateral implantation of the Vivity IOL (DAT***/CCWET*) performed by 4 surgeons using similar surgical techniques. 40 subjects will be enrolled.

Patients will be assessed for monocular and binocular distance, intermediate, and near vision.

The hypothesis is that post-refractive patients that have high spherical aberration (SAs) will have excellent outcomes and satisfaction with a Vivity IOL

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 40 years of age having already undergone cataract removal by phacoemulsification with a clear corneal incision in both eyes with implantation of the Vivity IOL (DAT***/CCWET*)
2. Prior uncomplicated, distance-targeted, bilateral myopic LASIK or PRK (photorefractive keratectomy) surgery and corneal spherical aberration greater than ≥0.30 μ and ≤ 1.20 μ in at least one eye (6.00 mm) as measured at their cataract pre-op visit
3. Able to comprehend and willing to sign informed consent and complete all required testing procedures
4. Best Corrected Distance Visual Acuity (BCDVA) projected to be 0.10 logMAR (Minimum Angle of Resolution) or better
5. Clear intraocular media
6. Minimum of two weeks post YAG (yttrium aluminum garnet) capsulotomy to treat PCO (posterior capsular opacification)
7. Residual refractive astigmatism ≤0.50 diopters
8. Post-operative refractive spherical equivalent from +0.50 to -0.50 spherical equivalent

Exclusion Criteria:

1. Any corneal abnormality, other than regular corneal astigmatism or myopic LASIK/PRK surgery, (as determined by pre-operative testing) that in the opinion of the investigator would confound the outcome(s) of the study
2. Any complication during cataract surgery (capsular tear, vitrectomy, etc)
3. History of or current retinal conditions or predisposition to retinal conditions or predisposition to retinal conditions
4. Amblyopia or strabismus in either eye
5. History of or current anterior or posterior segment inflammation of any etiology
6. Any form of neovascularization on or within the eye
7. Glaucoma (uncontrolled or controlled with medication)
8. Optic nerve atrophy
9. Subjects with diagnosed degenerative eye disorders
10. Postoperative CDVA worse than 0.10 logMAR in either eye.
11. Subjects who have an acute or chronic disease or illness that would confound the results of this investigation in the opinion of the principal investigator (e.g. immunocompromised, connective tissue disease, clinically significant atopic disease, etc)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with healthy eyes, prior myopic LASIK or PRK with SA greater than 0.3, and uncomplicated bilateral implantation of the Vivity IOL (DAT***/CCWET*).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Micheletti, MD, Principal Investigator — Berkeley Eye Center
Locations (1):
- Berkeley Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Vivity IOL Group
Started | 20; 40 eyes
Completed | 20; 40 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Binocular Best Corrected Distance Visual Acuity
Description: Binocular Best Corrected Distance Visual Acuity in logMAR
Time Frame: 3 weeks post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
logMAR | -0.05 (0.09)

2. Secondary Outcome: Monocular Visual Acuity
Description: Monocular UDVA (uncorrected distance visual acuity), UIVA (uncorrected intermediate visual acuity), UNVA (uncorrected near visual acuity), and CDVA (corrected distance visual acuity)
Time Frame: 3 weeks post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
Number analyzed (eyes) | 40
logMAR
  UDVA | 0.06 (0.11)
  UIVA | 0.18 (0.12)
  UNVA | 0.31 (0.19)
  CDVA | 0.00 (0.08)

3. Secondary Outcome: Binocular Distance, Intermediate, and Near Visual Acuity
Description: Binocular distance (UDVA), intermediate (UIVA, DCIVA), and near visual acuity (UNVA, DCNVA)
Time Frame: 3 weeks post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
logMAR
  UDVA | 0.02 (0.16)
  UIVA | 0.14 (0.13)
  DCIVA | 0.11 (0.11)
  UNVA | 0.24 (0.14)
  DCNVA | 0.25 (0.15)

4. Secondary Outcome: Quality of Vision After Surgery (QUVID) Questionnaire
Description: Patient reported disphotopsias by QUVID questionnaire will be assessed. Variables measured on a categorical scale will be summarized to provide the number and percentage of subjects who provided each score. The percentage of subjects that answered "Never" or "Rarely" for frequency are provided.
Time Frame: 3 weeks post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
Participants
  Starburst | 11
  Halos | 13
  Glare | 9
  Haze | 15
  Blurred Vision | 15
  Double Vision | 19
  Dark Area | 20

5. Secondary Outcome: Intraocular Lens Satisfaction (IOLSAT) Questionnaire
Description: Patient reported satisfaction by IOLSAT questionnaire will be assessed. Variables measured on a categorical scale will be summarized to provide the number and percentage of subjects who provided each score. The percentage of patients "Satisfied" or "Very Satisfied" will be added for a total satisfaction percentage.
Time Frame: 3 weeks post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
Participants | 16

6. Secondary Outcome: Post-op Refraction
Description: Manifest refraction spherical equivalent (MRSE)
Time Frame: 3 weeks post operatively
Measure: Mean (Standard Deviation); unit: D
Units Other Than Participants: eyes
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
Number analyzed (eyes) | 40
D | -0.11 (0.31)

7. Other Pre Specified Outcome: Binocular Defocus Curve
Description: Binocular defocus curve (distance corrected)
Time Frame: 3 weeks post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
logMAR
  -3.00 D | 0.39 (0.17)
  -2.50 D | 0.26 (0.17)
  -2.00 D | 0.17 (0.13)
  -1.50 D | 0.05 (0.12)
  -1.00 D | 0.03 (0.11)
  -0.50 D | 0.00 (0.11)
  -0.25 D | -0.05 (0.09)
  0.00 D | -0.06 (0.09)
  0.25 D | -0.02 (0.10)
  0.50 D | 0.00 (0.10)
  1.00 D | 0.11 (0.10)

8. Other Pre Specified Outcome: Spectacle Independence (IOLSAT)
Description: Spectacle independence utilizing the IOLSAT will be assessed. Variables measured on a categorical scale will be summarized to provide the number and percentage of subjects who provided each score. Spectacle independence was defined as answering "Never" or "Rarely" on the IOLSAT, the data presented is the percentage of subjects answering "Never" or "Rarely".
Time Frame: 3 weeks post operatively
Measure: Number; unit: percentage of participants
Arm/Group | Vivity IOL Group
Number analyzed (Participants) | 20
percentage of participants
  Overall | 90
  Distance | 90
  Intermediate | 75
  Near | 30

ADVERSE EVENTS:
Time Frame: 3 weeks postoperatively
Arm/Group | Vivity IOL Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT06064916/Prot_000.pdf